CLINICAL TRIAL: NCT03133546
Title: A Randomised Phase II Trial of Osimertinib and Bevacizumab Versus Osimertinib Alone as Second-line Treatment in Stage IIIb-IVb NSCLC With Confirmed EGFRm and T790M
Brief Title: Osimertinib and Bevacizumab Versus Osimertinib Alone as Second-line Treatment in Stage IIIb-IVb NSCLC With Confirmed EGFRm and T790M
Acronym: BOOSTER
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ETOP IBCSG Partners Foundation (Network)
Collaborators: AstraZeneca (Industry); Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ETOP 10-16; 2016-002029-12 (EudraCT Number); ESR-15-11666 (Other: AstraZeneca); MO39447 (Other: Roche)
Record Dates: First submitted 2017-04-20; First posted 2017-04-28 (Actual); Results first posted 2025-01-14 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2025-01

CONDITIONS: Non Small Cell Lung Cancer Metastatic
Keywords: NSCLC; EGFR; TKI; EGFRm; T790M
MeSH Terms: interventions — osimertinib; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Osimertinib plus Bevacizumab (Experimental): Patients will receive treatment with osimertinib and bevacizumab until disease progression, lack of tolerability or the patient declines further treatment. Treatment may also continue beyond progression for as long as the patient may still derive benefit.
  Interventions: Drug: Osimertinib; Drug: Bevacizumab
- Osimertinib alone (Active Comparator): Patients will receive treatment with osimertinib until disease progression, lack of tolerability or the patient declines further treatment. Treatment may also continue beyond progression for as long as the patient may still derive benefit.
  Interventions: Drug: Osimertinib

INTERVENTIONS:
Drug: Osimertinib — Osimertinib is administered orally at 80mg once daily. Doses should be taken approximately 24 hours apart at the same time point each day. The appropriate number of osimertinib tablets will be provided to patients to be self-administered at home. AstraZeneca will supply osimertinib as tablets for oral administration.
  AstraZeneca will supply osimertinib as tablets for oral administration.
  Other Names: Tagrisso
Drug: Bevacizumab — Bevacizumab is administered at 15mg/kg intravenously on day 1 of every 3-week cycle. Bevacizumab for intravenous administration will be supplied by Roche.
  Other Names: Avastin
  Arms: Osimertinib plus Bevacizumab

SUMMARY:
BOOSTER is a randomised, controlled, phase II trial comparing osimertinib and bevacizumab versus osimertinib alone as second-line treatment in patients with stage IIIb-IVb non-small cell lung carcinoma (NSCLC) harbouring activating EGFR (exon 19 deletion or L858R) and T790M resistance mutation.

DETAILED DESCRIPTION:
Lung cancer has been the most common carcinoma in the world for several decades. Non-small cell lung carcinoma (NSCLC) represents approximately 80-85% of all lung cancers. At the time of diagnosis approximately 70% of NSCLC patients already have advanced or metastatic disease not amenable to surgical resection. A significant percentage of early stage NSCLC patients who have undergone surgery subsequently develop distant recurrence.

First-generation EGFR tyrosine kinase inhibitors (TKIs) provide significant clinical benefit in patients with advanced EGFR-mutant (EGFRm) non-small cell lung carcinoma (NSCLC). However, all patients ultimately develop disease progression, driven - as the most prevalent identified biological mechanism - by the acquisition of a second T790M EGFR TKI resistance mutation.

Osimertinib (AZD9291) is a novel oral, potent, and selective third-generation irreversible inhibitor of both EGFRm-sensitizing and T790M resistance mutants. This mono-anilino-pyrimidine compound is structurally distinct from other third-generation EGFR TKIs and offers a pharmacologically differentiated profile from earlier first and second generation EGFR TKIs.

Osimertinib is being evaluated in several prospective clinical trials, notably in frontline treatment, in the adjuvant setting, and in combination with later lines in EGFRm positive advanced disease. Combination treatments that target both tumour cells and tumour microenvironment (such as angiogenesis) may be a promising strategy for further improving efficacy outcomes in patients with EGFRm NSCLC following progression on EGFR TKI therapy and other lines of therapy. There is thus a considerable unmet clinical need for novel therapeutic options that can further extend the efficacy of targeted agents such as EGFR TKIs, across all lines of therapy.

Bevacizumab is a recombinant humanized monoclonal IgG1 antibody that binds to and inhibits the interaction of VEGF-A to its receptors (Flt-1 and KDR) on the surface of endothelial cells. The interaction of VEGF with its receptors leads to endothelial cell proliferation and new blood vessel formation in in vitro models of angiogenesis. Neutralising the biological activity of VEGF regresses the vascularisation of tumours, normalises remaining tumour vasculature, and inhibits the formation of new tumour vasculature, thereby inhibiting tumour growth. Bevacizumab is indicated for the first-line treatment of unresectable, locally advanced, recurrent or metastatic non-squamous NSCLC in combination with carboplatin and paclitaxel.

Osimertinib monotherapy, at the dose to be evaluated in this trial, has shown consistent and high objective response rates in the target patient population.

Anti-angiogenic agents targeting the VEGF/VEGFR signalling pathway have been shown to provide additional efficacy when used in combination with first-line platinum-based chemotherapy in several trials in non-squamous NSCLC or in combination with erlotinib as first line therapy in EGFRm positive NSCLC patients. The combination of osimertinib plus an anti-angiogenic agent such as bevacizumab may provide a wider activity against tumours that have developed resistance to EGFR TKI agents by blocking the dual pathways of proliferative signalling and antigenic signalling. Preclinical studies suggested that patients on lower doses of EGFR TKI tend to develop treatment resistance earlier than those who receive higher doses. Therefore the combination may also delay the development of subsequent resistance as the preclinical studies suggested anti-angiogenic agents may increase intratumoural uptake of anti-cancer drugs by changing tumour vessel physiology.

Efficacy and safety data from the osimertinib monotherapy studies have shown promising efficacy and an acceptable safety profile at the recommended dose of 80 mg once daily. The combination of osimertinib with bevacizumab may have the potential to provide additional clinical benefit in terms of increased and/or prolonged disease control and a delay in the emergence of resistance in patients with advanced EGFRm NSCLC who have progressed following a prior EGFR TKI agent, compared against the current standard of care (chemotherapy or another EGFR TKI) or monotherapy of any of the individual agents.

ELIGIBILITY:
Inclusion Criteria:

* Patients (male/female) must be >18 years of age.
* Patients diagnosed with NSCLC, stage IIIb/IIIc (not amenable to radical therapy) or IVa/IVb according to 8th TNM classification, after progression following prior EGFR TKI therapy (erlotinib, gefitinib, dacomitinib or afatinib) as the most recent treatment regimen;
* Pathological diagnosis of predominantly non-squamous NSCLC;
* Maximum one line of previous platinum based chemotherapy;
* Histological or cytological confirmation of EGFRm (exon 19 deletion or exon 21L858R);
* Locally confirmed T790M mutation determined from biopsy (preferred) or on circulating tumour DNA, documented in tissue, plasma or serum after disease progression on the most recent treatment regimen;
* Plasma, serum, and tumour (preferred) tissue or cytology (if biopsy was taken and FFPE tumor material is not yet fully depleted) after disease progression on the most recent EGFR TKI treatment available for central confirmation of T790M;
* Measurable or evaluable disease according to RECIST 1.1;
* Adequate haematological, renal and liver function;
* World Health Organization (WHO) performance status 0-2.

Exclusion Criteria:

* Patients with mixed NSCLC with predominantly squamous cell cancer, or with any small cell lung cancer (SCLC) component;
* Symptomatic or active central nervous system metastases, as indicated by progressive growth or increasing need of steroids.
* Patients currently receiving medications or herbal supplements known to be potent CYP3A4 inducers;
* Patients with any unresolved toxicities from prior therapy greater than CTCAE V 4.0 grade 1 (exception: alopecia & grade 2, prior platinuma-therapy related neuropathy)
* Previous treatment with osimertinib and/or bevacizumab;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2017-05-31 (Actual); Primary Completion 2021-02-22 (Actual); Study Completion 2024-02-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Solange Peters, MD, Study Chair — Centre Hospitalier Universitaire Vaudois; Rolf Stahel, MD, Study Chair — University Hospital Zuerich, Zurich, Switzerland
Locations (25):
- Ireland (2):
  - St. James Hospital, Dublin
  - Mid Western Cancer Centre, Limerick
- VU University Medical Centre, Amsterdam, Netherlands
- Singapore (2):
  - National University Hospital, Singapore
  - Tan Tock Seng Hospital, Singapore
- South Korea (2):
  - National Cancer Centre, Goyang
  - Severance Hospital, Yonsei University Health System, Seoul
- Spain (13):
  - Hospital Teresa Herrara, A Coruña
  - Hospital General Alicante, Alicante
  - Hospital Sant Pau, Barcelona
  - ICO Badalona, Barcelona
  - ICO Hospitalet, Barcelona
  - OSI Bilbao Basurto, Bilbao
  - Fund. Jimenez Diaz, Madrid
  - Hospital de la Princesa, Madrid
  - Hospital la Paz, Madrid
  - Hospital Puerta de Hierro, Madrid
  - Hospital Virgen del Rocio, Seville
  - Hospital Arnau de Vilanova, Valencia
  - Hospital General de Valencia, Valencia
- Switzerland (5):
  - Geneva University Hospital (HUG), Geneva
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - Kantonsspital St. Gallen, Sankt Gallen
  - Kantonsspital Winterthur, Winterthur
  - UniversitatSpital Zurich, Zurich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bonomi PD. Implications of key trials in advanced nonsmall cell lung cancer. Cancer. 2010 Mar 1;116(5):1155-64. doi: 10.1002/cncr.24815. PMID 20087963
- [Background] Jackman DM, Miller VA, Cioffredi LA, Yeap BY, Janne PA, Riely GJ, Ruiz MG, Giaccone G, Sequist LV, Johnson BE. Impact of epidermal growth factor receptor and KRAS mutations on clinical outcomes in previously untreated non-small cell lung cancer patients: results of an online tumor registry of clinical trials. Clin Cancer Res. 2009 Aug 15;15(16):5267-73. doi: 10.1158/1078-0432.CCR-09-0888. Epub 2009 Aug 11. PMID 19671843
- [Background] Oxnard GR, Arcila ME, Sima CS, Riely GJ, Chmielecki J, Kris MG, Pao W, Ladanyi M, Miller VA. Acquired resistance to EGFR tyrosine kinase inhibitors in EGFR-mutant lung cancer: distinct natural history of patients with tumors harboring the T790M mutation. Clin Cancer Res. 2011 Mar 15;17(6):1616-22. doi: 10.1158/1078-0432.CCR-10-2692. Epub 2010 Dec 6. PMID 21135146
- [Background] Rosell R, Carcereny E, Gervais R, Vergnenegre A, Massuti B, Felip E, Palmero R, Garcia-Gomez R, Pallares C, Sanchez JM, Porta R, Cobo M, Garrido P, Longo F, Moran T, Insa A, De Marinis F, Corre R, Bover I, Illiano A, Dansin E, de Castro J, Milella M, Reguart N, Altavilla G, Jimenez U, Provencio M, Moreno MA, Terrasa J, Munoz-Langa J, Valdivia J, Isla D, Domine M, Molinier O, Mazieres J, Baize N, Garcia-Campelo R, Robinet G, Rodriguez-Abreu D, Lopez-Vivanco G, Gebbia V, Ferrera-Delgado L, Bombaron P, Bernabe R, Bearz A, Artal A, Cortesi E, Rolfo C, Sanchez-Ronco M, Drozdowskyj A, Queralt C, de Aguirre I, Ramirez JL, Sanchez JJ, Molina MA, Taron M, Paz-Ares L; Spanish Lung Cancer Group in collaboration with Groupe Francais de Pneumo-Cancerologie and Associazione Italiana Oncologia Toracica. Erlotinib versus standard chemotherapy as first-line treatment for European patients with advanced EGFR mutation-positive non-small-cell lung cancer (EURTAC): a multicentre, open-label, randomised phase 3 trial. Lancet Oncol. 2012 Mar;13(3):239-46. doi: 10.1016/S1470-2045(11)70393-X. Epub 2012 Jan 26. PMID 22285168
- [Background] Finlay MR, Anderton M, Ashton S, Ballard P, Bethel PA, Box MR, Bradbury RH, Brown SJ, Butterworth S, Campbell A, Chorley C, Colclough N, Cross DA, Currie GS, Grist M, Hassall L, Hill GB, James D, James M, Kemmitt P, Klinowska T, Lamont G, Lamont SG, Martin N, McFarland HL, Mellor MJ, Orme JP, Perkins D, Perkins P, Richmond G, Smith P, Ward RA, Waring MJ, Whittaker D, Wells S, Wrigley GL. Discovery of a potent and selective EGFR inhibitor (AZD9291) of both sensitizing and T790M resistance mutations that spares the wild type form of the receptor. J Med Chem. 2014 Oct 23;57(20):8249-67. doi: 10.1021/jm500973a. Epub 2014 Oct 1. PMID 25271963
- [Background] Camidge DR, Pao W, Sequist LV. Acquired resistance to TKIs in solid tumours: learning from lung cancer. Nat Rev Clin Oncol. 2014 Aug;11(8):473-81. doi: 10.1038/nrclinonc.2014.104. Epub 2014 Jul 1. PMID 24981256

RESULTS

PARTICIPANT FLOW:
Groups:
- Osimertinib Plus Bevacizumab: Patients will receive treatment with osimertinib and bevacizumab until disease progression, lack of tolerability or the patient declines further treatment. Treatment may also continue beyond progression for as long as the patient may still derive benefit.
  Osimertinib: Osimertinib is administered orally at 80mg once daily. Doses should be taken approximately 24 hours apart at the same time point each day. The appropriate number of osimertinib tablets will be provided to patients to be self-administered at home. AstraZeneca will supply osimertinib as tablets for oral administration.
  AstraZeneca will supply osimertinib as tablets for oral administration.
  Bevacizumab: Bevacizumab is administered at 15mg/kg intravenously on day 1 of every 3-week cycle. Bevacizumab for intravenous administration will be supplied by Roche.
- Osimertinib Alone: Patients will receive treatment with osimertinib until disease progression, lack of tolerability or the patient declines further treatment. Treatment may also continue beyond progression for as long as the patient may still derive benefit.
  Osimertinib: Osimertinib is administered orally at 80mg once daily. Doses should be taken approximately 24 hours apart at the same time point each day. The appropriate number of osimertinib tablets will be provided to patients to be self-administered at home. AstraZeneca will supply osimertinib as tablets for oral administration.
  AstraZeneca will supply osimertinib as tablets for oral administration.
Period: Overall Study
Arm/Group | Osimertinib Plus Bevacizumab | Osimertinib Alone
Started | 78 | 77
Received at least one dose of trial treatment (Safety cohort: patients at risk for adverse events and serious adverse events) | 76 | 77
On treatment (At database cut-off for final efficacy analysis: February 22, 2021) | 1 | 8
Treatment failures (Osimertinib plus Bevacizumab: 36 toxicities, 29 progressions, 4 other reasons, 3 patient decisions, 2 deaths, 1 investigator decision Osimertinib alone: 3 toxicities, 53 progressions, 1 other reason, 4 patient decisions, 7 deaths, 1 investigator decision) | 75 | 69
Never started treatment | 2 | 0
Completed (Still on follow-up at database cut-off for final efficacy analysis: February 22, 2021) | 27 | 27
Not Completed | 51 | 50
Not completed — Death | 46 | 43
Not completed — Withdrawal/Lost to follow-up | 5 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Osimertinib Plus Bevacizumab | Osimertinib Alone | Total
Number analyzed (Participants) | 78 | 77 | 155
Age, Continuous [Median (Full Range); unit: years] | 68 [34 to 85] | 66 [41 to 83] | 67 [34 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 49 | 96
  Male | 31 | 28 | 59
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 32 | 31 | 63
  Non-Asian | 46 | 46 | 92
ECOG Performance Status [Count of Participants; unit: Participants] — 0: Fully active, able to carry on all pre-disease performance without restriction; 1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work; 2: Ambulatory and capable of all selfcare but unable to carry out any work activities, up and about more than 50% of waking hours.
  Participants
    0 | 22 | 25 | 47
    1 | 51 | 48 | 99
    2 | 5 | 4 | 9
Smoking status [Count of Participants; unit: Participants] — Current smoker: Still smokes cigarettes, Former smoker: Smoked at least 100 cigarettes in the past during the whole life, Never smoker: Smoked 0-99 cigarettes during the whole life.
  Participants
    Current smoker | 4 | 1 | 5
    Former smoker | 30 | 27 | 57
    Never smoked | 44 | 49 | 93
Stage [Count of Participants; unit: Participants] — Stage is based on the 8th TNM classification for NSCLC (American Joint Committee on Cancer).
  Stage IIIB/C: the tumor is 5 cm or smaller (IIIB) or any size (IIIC) and cancer has spread to lymph nodes above the collarbone on the same side of the chest as the primary tumor or to any lymph nodes on the opposite side of the chest as the primary tumor.
  Stage IVA: cancer has spread within the chest and/or has spread to 1 area outside of the chest.
  Stage IVB: cancer has spread outside of the chest to more than 1 place in 1 organ or to more than 1 organ.
  Participants
    IIIB/C | 2 | 0 | 2
    IVA/B | 76 | 76 | 152
    Missing | 0 | 1 | 1
Use of prior platinum-based chemotherapy [Count of Participants; unit: Participants] | 11 | 13 | 24
Prior EGFR TKI [Count of Participants; unit: Participants] — TKI: tyrosine kinase inhibitors
  Participants
    Erlotinib/gefitinib | 57 | 57 | 114
    Afatinib/dacomitinib | 21 | 19 | 40
    Other | 0 | 1 | 1
EGFR mutation type [Count of Participants; unit: Participants] — Histologically or cytologically confirmed exon 19 deletion or exon 21 L858R mutation by a certified local laboratory
  Participants
    Exon 19 deletion | 58 | 51 | 109
    Exon 21 L858R | 20 | 26 | 46
T790M testing material [Count of Participants; unit: Participants] — Confirmation of T790M mutation determined from biopsy or on serum circulating tumour DNA by a certified local laboratory. These samples must be taken after disease progression on the most recent EGFR TKI regimen.
  Participants
    ctDNA | 38 | 37 | 75
    Tumour | 40 | 40 | 80
Brain metastasis [Count of Participants; unit: Participants]
  Yes | 13 | 8 | 21
  No | 65 | 69 | 134
Liver metastasis [Count of Participants; unit: Participants]
  Yes | 14 | 8 | 22
  No | 64 | 69 | 133
Pleural effusion and ascites [Count of Participants; unit: Participants]
  Yes | 7 | 9 | 16
  No | 71 | 68 | 139

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the time from the date of randomisation until documented progression (based on RECIST 1.1 criteria) or death, if progression is not documented. Censoring (for patients without progression/death) will occur at the last tumour assessment if patient is lost to follow-up or refuses further documentation of follow-up.
Time Frame: Evaluated up to approximately 45 months from the randomisation of the first patient.
Population: Efficacy population (Intention-To-Treat cohort of all randomised patients)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Osimertinib Plus Bevacizumab | Osimertinib Alone
Number analyzed (Participants) | 78 | 77
months | 15.4 [9.2 to 18] | 12.3 [6.2 to 17.2]
Statistical Analysis 1: Comparison: Osimertinib Plus Bevacizumab vs Osimertinib Alone; Assumption: Median PFS with osimertinib 11 months Target: Detect a 36% improvement in PFS (HR=0.64, corresponding to an increase in median PFS to 17.2 months) under osimertinib and bevacizumab (80% power, at one-sided significant level of 5%) 126 events required; Test type: Superiority; p = 0.84, Regression, Cox — significance level: 5%; Univariate Cox for PFS with treatment effect only; Hazard Ratio (HR) = 0.96, 95% CI 2-sided [0.68 to 1.37] — The HR for Osimertinib plus Bevacizumab versus Osimertinib alone is provided

2. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR is defined as the percentage of patients reaching a complete or partial response, across all assessment time-points according to RECIST criteria v1.1, during the period from randomisation to termination of trial treatment.
Time Frame: Evaluated up to approximately 45 months from the randomisation of the first patient.
Population: Efficacy population (Intention-To-Treat cohort of all randomised patients)
Measure: Count of Participants; unit: Participants
Arm/Group | Osimertinib Plus Bevacizumab | Osimertinib Alone
Number analyzed (Participants) | 78 | 77
Participants | 43 | 42

3. Secondary Outcome: Disease Control Rate (DCR)
Description: DCR is defined as the percentage of patients reaching a complete or partial response, or disease stabilisation confirmed at subsequent radiological assessment, across all assessment time-points according to RECIST criteria v1.1, during the period from randomisation to termination of trial treatment.
Time Frame: Evaluated up to approximately 45 months from the randomisation of the first patient.
Population: Efficacy population (Intention-To-Treat cohort of all randomised patients)
Measure: Count of Participants; unit: Participants
Arm/Group | Osimertinib Plus Bevacizumab | Osimertinib Alone
Number analyzed (Participants) | 78 | 77
Participants | 70 | 63

4. Secondary Outcome: Adverse Events
Description: Adverse events, graded by CTCAE version 4.0, will be recorded from date of signature of informed consent until 30 days after all trial treatment discontinuation.
Time Frame: Evaluated up to approximately 45 months from the randomisation of the first patient.
Population: Safety population (all patients who received at least 1 dose of trial treatment).
Measure: Count of Participants; unit: Participants
Arm/Group | Osimertinib Plus Bevacizumab | Osimertinib Alone
Number analyzed (Participants) | 76 | 77
Participants
  Experienced AE/SAE | 76 | 76
  No AE/SAE | 0 | 1
  Experienced SAE | 33 | 27

5. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as time from the date of randomisation until death from any cause. Censoring will occur at the last follow-up date.
Time Frame: Evaluated up to approximately 45 months from the randomisation of the first patient.
Population: Efficacy population (Intention-To-Treat cohort of all randomised patients)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Osimertinib Plus Bevacizumab | Osimertinib Alone
Number analyzed (Participants) | 78 | 77
months | 24.0 [17.8 to 32.1] | 24.3 [16.9 to 37.0]

6. Other Pre Specified Outcome: T790M Evolution in Tissue and Plasma/Serum Between Baseline and Disease Progression (PD) on Trial Treatment.
Description: Tumour tissue blocks, plasma and serum samples will be collected at trial entry and at disease progression on trial treatment.
Time Frame: Available for translational research, following completion of the primary trial research objectives.
Population: Patients with available NGS plasma sample.
Measure: Count of Participants; unit: Participants
Arm/Group | Osimertinib Plus Bevacizumab | Osimertinib Alone
Number analyzed (Participants) | 76 | 73
Participants
  T790M base to PD: No clearance | 8 | 8
  T790M base to PD: Clearance | 18 | 13
  T790M base to PD: Mutation at PD only | 0 | 1
  T790M base to PD: No mutation | 6 | 8
  T790M base to PD: Missing | 22 | 25
  T790M base to PD: Not applicable (No PD) | 22 | 18

ADVERSE EVENTS:
Time Frame: Continuously from date of Informed Consent signature until 30 days after all treatments discontinuation, up to approximately 45 months from the randomisation of the first patient.
Description: Adverse event (AE) is defined as any untoward medical occurrence that occurs from the date of signature of informed consent until 30 days after all trial treatment discontinuation, regardless of whether it is considered related to a medication. Adverse events are classified according to CTCAE version 4.0.
Arm/Group | Osimertinib Plus Bevacizumab | Osimertinib Alone
All-Cause Mortality (participants affected / at risk) | 46/78 | 43/77
Serious Adverse Events (participants affected / at risk) | 33/76 | 27/77
Other Adverse Events (participants affected / at risk) | 76/76 | 76/77
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Osimertinib Plus Bevacizumab (N=76) | Osimertinib Alone (N=77)
Diarrhea (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Mucositis oral (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 3
Abdominal pain (Gastrointestinal disorders) | 0 | 2
Gastrointestinal pain (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Gastric perforation (Gastrointestinal disorders) | 1 | 0
Lipase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Laryngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Splenic infection (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Fever (General disorders) | 0 | 2
Drug overdose (General disorders) | 3 | 2
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 | 0
Upper respiratory infection (Infections and infestations) | 1 | 2
Urinary tract infection (Infections and infestations) | 2 | 0
Lung infection (Infections and infestations) | 4 | 2
Pharyngitis (Infections and infestations) | 0 | 1
Bronchial infection (Infections and infestations) | 1 | 0
COVID-19 infection (Infections and infestations) | 1 | 0
Enterocolitis infectious (Infections and infestations) | 1 | 0
Hepatitis caused by COVID-19 infection (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Influenza A (Infections and infestations) | 1 | 0
Necrotising fasciitis (Infections and infestations) | 0 | 1
Pleural infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 | 0
Seizure (Nervous system disorders) | 1 | 1
Depressed level of consciousness (Nervous system disorders) | 1 | 0
Ischemia cerebrovascular (Nervous system disorders) | 1 | 0
Stroke (Nervous system disorders) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Thromboembolic event (Vascular disorders) | 2 | 3
Hematuria (Renal and urinary disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Mania (Psychiatric disorders) | 0 | 1
Heart failure (Cardiac disorders) | 2 | 0
Atrial fibrillation (Cardiac disorders) | 3 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1
Pleurodesis of malignant pleural effusion (Surgical and medical procedures) | 0 | 1
Fracture (Injury, poisoning and procedural complications) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 1
Autoimmune disorder (Immune system disorders) | 0 | 1
Gastric carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Osimertinib Plus Bevacizumab (N=76) | Osimertinib Alone (N=77)
Diarrhea (Gastrointestinal disorders) | 41 | 38
Constipation (Gastrointestinal disorders) | 19 | 16
Mucositis oral (Gastrointestinal disorders) | 19 | 10
Nausea (Gastrointestinal disorders) | 17 | 13
Vomiting (Gastrointestinal disorders) | 17 | 7
Abdominal pain (Gastrointestinal disorders) | 7 | 4
Dry mouth (Gastrointestinal disorders) | 2 | 8
Lipase increased (Investigations) | 12 | 13
Serum amylase increased (Investigations) | 12 | 13
Platelet count decreased (Investigations) | 15 | 9
Neutrophil count decreased (Investigations) | 7 | 10
Alanine aminotransferase increased (Investigations) | 10 | 6
Aspartate aminotransferase increased (Investigations) | 10 | 5
Electrocardiogram QT corrected interval prolonged (Investigations) | 10 | 5
Ejection fraction decreased (Investigations) | 9 | 1
Alkaline phosphatase increased (Investigations) | 6 | 3
Creatinine increased (Investigations) | 7 | 2
White blood cell decreased (Investigations) | 5 | 4
GGT increased (Investigations) | 6 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 31 | 28
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 13 | 17
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 16 | 4
Sore throat (Respiratory, thoracic and mediastinal disorders) | 7 | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 5
Rash acneiform (Skin and subcutaneous tissue disorders) | 27 | 19
Dry skin (Skin and subcutaneous tissue disorders) | 16 | 15
Pruritus (Skin and subcutaneous tissue disorders) | 8 | 15
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 6 | 5
Upper respiratory infection (Infections and infestations) | 16 | 15
Paronychia (Infections and infestations) | 13 | 13
Urinary tract infection (Infections and infestations) | 6 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 10 | 11
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 9
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 3
Headache (Nervous system disorders) | 18 | 9
Dizziness (Nervous system disorders) | 9 | 11
Anorexia (Metabolism and nutrition disorders) | 24 | 17
Hyponatremia (Metabolism and nutrition disorders) | 6 | 4
Hypokalemia (Metabolism and nutrition disorders) | 3 | 6
Hypertension (Vascular disorders) | 32 | 7
Proteinuria (Renal and urinary disorders) | 37 | 2
Dry eye (Eye disorders) | 4 | 10
Blurred vision (Eye disorders) | 4 | 5
Anxiety (Psychiatric disorders) | 1 | 7
Anemia (Blood and lymphatic system disorders) | 7 | 12
Fatigue (General disorders) | 33 | 29
Pain (General disorders) | 22 | 12
Fever (General disorders) | 6 | 10
Edema limbs (General disorders) | 10 | 4
Non-cardiac chest pain (General disorders) | 9 | 1
Flu like symptoms (General disorders) | 6 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-11-14): https://cdn.clinicaltrials.gov/large-docs/46/NCT03133546/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-23): https://cdn.clinicaltrials.gov/large-docs/46/NCT03133546/SAP_001.pdf